CLINICAL TRIAL: NCT06213467
Title: Pain Perception and Evaluated Injectable Anesthesia Needed by Using Pulsating Diode Laser 940nm in Second Stage Implant Exposure Versus Traditional Methods
Brief Title: Using Diode Laser in 2nd Stage of Implant.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Baghdad (Other)
Responsible Party: Principal Investigator, Saad Mahmood Jameel, Msc student, University of Baghdad
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1375
Record Dates: First submitted 2024-01-09; First posted 2024-01-19 (Actual); Last update posted 2024-01-19 (Actual); Status verified 2024-01

CONDITIONS: Dental Implant Exposure Using Diode Laser
Keywords: diode laser; dental implant; local anasthesia
MeSH Terms: interventions — Lasers, Semiconductor

STUDY DESIGN:
Intervention Model Description: 15 patients that have at least two dental implants in jaws.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- A and B (Experimental): Each patient in which two implants have already been inserted are exposed, the first implant expose by using traditional methods , the second one expose by using diode laser 940nm .
  Interventions: Device: diode laser 940nm

INTERVENTIONS:
Device: diode laser 940nm — Exposure for the two implants was done at the same visit, with one implant being exposed using diode laser and the other implant using traditional method

SUMMARY:
Dental Implants that are teeth replacements usually place with two stages. In the second stage the implant fixture, (which is the body that inserted in the bone is exposed to place the artificial tooth), is exposed using surgical blade, however; an alternative method using diode laser may be used. This study aimed to compare the two methods in relation to pain anticipated by the patients and the need for local anesthesia usage.

DETAILED DESCRIPTION:
Second-stage implant exposure involves removing soft tissue above the dental implant, as a part of the implant procedures to replace the missing teeth which can be done either by using diode laser or traditional method This study included fifteen patients, aged between 18 and 70 years old. Implant exposure was performed on 15 patients has at least two implants in two groups: group 1 with a diode laser at 940nm and group 2 with the traditional method performed either using a puncture, flap, or incision in 5 private clinics and one governmental run hospital in city of Baghdad/ Iraq.

ELIGIBILITY:
Inclusion Criteria:

- 1. Describe the target population and the criteria for their inclusion. Patients indicated for fixed implant treatment with conventional Implant procedure with implant insertd before (3-6) months by using two stage dental implant.

2. Treatment with two or more implant in same patient. 3. Patients aged from 18 to 70 years of both the gender with the presence of adequate osseointegration and healthy keratinized tissue surrounding the implant site.

Exclusion Criteria:

* 1. Patient have single implant. 2. Expose dental implant or already have gingival former. 3. Poor oral hygiene. 4. Failure implant osseointegration to bone.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2022-11-21 (Actual); Primary Completion 2023-11-16 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Pain perceived by the patient. | recordings were done immediately at time of exposure , after 2 , 5 ,7 days postsurgical.
  Pain was measured using visual analogue scale from 0-10, filled by the patient

SECONDARY OUTCOMES:
need for injectable anesthesia | at time of operation treatment
  need for anesthesia done when patient feels pain after application of local anesthesia

CONTACTS AND LOCATIONS:
Locations (1):
- laser institute for postgraduate studies, University of Baghdad, Baghdad, Al-Jadiriya, Iraq

IPD SHARING:
Plan to Share IPD: No
will be provided when needed